CLINICAL TRIAL: NCT01852539
Title: Optimal Dose of Dexmedetomidine for Laryngeal Mask Airway Insertion During Propofol Induction
Brief Title: Dexmedetomidine for Laryngeal Mask Airway Insertion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Associate professor, Ajou University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AJIRB-MED-CT4-13-045
Record Dates: First submitted 2013-05-03; First posted 2013-05-13 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-04

CONDITIONS: Drug Usage
Keywords: LMA insertion; dexmedetomidine; propofol
MeSH Terms: interventions — Dexmedetomidine; Propofol; Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dexmedetomidine (Experimental): After intravenous infusion of dexmedetomidine for 2 min, propofol 2.0 mg/kg was administrated. And laryngeal mask airway device was inserted(LMA # 3,4).
  Interventions: Drug: dexmedetomidine; Drug: propofol; Device: laryngeal mask airway (LMA)

INTERVENTIONS:
Drug: dexmedetomidine — The dose of dexmedetomidine was determined by modified Dixon's up-and-down method, starting from 0.5 μg/kg (0.1 μg/kg as a step size).
  Other Names: precedex
Drug: propofol — Propofol 2.0 mg/kg was administrated
  Other Names: 2% fresofol
Device: laryngeal mask airway (LMA) — The insertion of laryngeal mask airway (LMA) was attempted, after confirming the loss of eyelash reflex,the bispectral index (BIS) score decreased below 60.

SUMMARY:
The investigators attempted to determine the optimal dose of dexmedetomidine required for the successful insertion of LMA during propofol induction without a neuromuscular blocking agent.

DETAILED DESCRIPTION:
After a predetermined bolus dose of dexmedetomidine was injected over 2 min, anesthesia was induced with propofol 2.0 mg/kg. After confirming the loss of eyelash reflex and the bispectral index (BIS) score decreased below 60, the insertion of LMA was attempted.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients undergoing general anesthesia for short elective surgery (<1 hr)

Exclusion Criteria:

* G-E reflux
* obesity (BMI>30)
* anticipated difficult airway

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2013-07; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
successful insertion of LMA | from baseline to 2 min after insertion of LMA (participants will be followed for the duration of anesthetic induction, an expected average of 10 min).
  the response of patients to the insertion of LMA (classified as either 'movement' or 'no movement') during infusion of dexmedetomidine and propofol.

CONTACTS AND LOCATIONS:
Overall Officials: Jong Yeop Kim, MD, Study Director — Ajou University School of Medicine
Locations (1):
- Ajou University School of Medicine, Suwon, South Korea

REFERENCES:
- [Result] Uzumcugil F, Canbay O, Celebi N, Karagoz AH, Ozgen S. Comparison of dexmedetomidine-propofol vs. fentanyl-propofol for laryngeal mask insertion. Eur J Anaesthesiol. 2008 Aug;25(8):675-80. doi: 10.1017/S0265021508004213. Epub 2008 Apr 10. PMID 18400141